CLINICAL TRIAL: NCT06651866
Title: Dose Escalation Study of Liposomal Mitoxantrone Hydrochloride Injection Combined With Decitabine and Cytarabine (D-CMG) for the Treatment of Elderly Newly Diagnosed Acute Myeloid Leukemia (AML) Patients
Brief Title: Dose-escalation Study of D-CMG Regimen for the Treatment of Elderly Newly Diagnosed AML Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Bing, Xu, Principal Investigator, The First Affiliated Hospital of Xiamen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMDYYYXYK-14
Record Dates: First submitted 2024-10-19; First posted 2024-10-22 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- D-CMG (Experimental): Liposomal mitoxantrone hydrochloride injection (Doxorubicin®): Used after dilution with 250mL of 5% glucose injection (50mg/mL), with an intravenous drip time of at least 60 minutes.
  * Level 1: 12mg/m2, IV drip, day 4;
  * Level 2: 18mg/m2, IV drip, day 4; Decitabine: 25mg, IV drip, days 1-3; Cytarabine: 10mg/m2, every 12 hours, IV drip, days 4-10; G-CSF: 300 ug, IV drip, days 1-5; Each cycle is 4 weeks, with a total of 2 cycles, and DLT is observed in the first cycle.
  Note: Patients who achieve CR (Complete Remission) and PR (Partial Remission) in the first cycle can continue with the original dose for one more cycle, and then the investigator decides whether to continue this regimen or choose another regimen for maintenance therapy; Patients with NR (No Remission) in the first cycle will be withdrawn from this study.
  Interventions: Drug: D-CMG

INTERVENTIONS:
Drug: D-CMG — Liposomal mitoxantrone hydrochloride injection (Doxorubicin®): Used after dilution with 250mL of 5% glucose injection (50mg/mL), with an intravenous drip time of at least 60 minutes.
  * Level 1: 12mg/m2, IV drip, day 4;
  * Level 2: 18mg/m2, IV drip, day 4; Decitabine: 25mg, IV drip, days 1-3; Cytarabine: 10mg/m2, every 12 hours, IV drip, days 4-10; G-CSF: 300 ug, IV drip, days 1-5; Each cycle is 4 weeks, with a total of 2 cycles, and DLT is observed in the first cycle.
  Note: Patients who achieve CR (Complete Remission) and PR (Partial Remission) in the first cycle can continue with the original dose for one more cycle, and then the investigator decides whether to continue this regimen or choose another regimen for maintenance therapy; Patients with NR (No Remission) in the first cycle will be withdrawn from this study.

SUMMARY:
to observe the dose-limiting toxicity (DLT) of liposomal mitoxantrone hydrochloride injection combined with cytarabine and decitabine in the initial treatment of acute myeloid leukemia (AML), to explore the maximum tolerated dose (MTD) of the combined D-CMG regimen, and to evaluate its safety and efficacy

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed acute myeloid leukemia (non-M3) that has not been previously treated and cannot receive standard cytarabine and anthracycline induction therapy due to age, comorbidities, or patient preference.
2. Aged 60-75 years, both male and female, with an expected survival time of more than 3 months.
3. Estimated creatinine clearance rate ≥ 30 mL/min.
4. AST and ALT ≤ 3.0 x ULN (unless considered due to leukemic organ involvement). Bilirubin ≤ 1.5 x ULN (unless considered due to leukemic organ involvement).
5. ECOG Performance Status ≤ 2.
6. Able to understand and voluntarily provide informed consent.

Exclusion Criteria:

1. Acute promyelocytic leukemia (APL) and low-risk cytogenetics, such as t(8;21), inv(16), or t(16;16).
2. Active central nervous system leukemia.
3. History of myeloproliferative neoplasms (MPN), including myelofibrosis, primary thrombocythemia, polycythemia vera, chronic myeloid leukemia (CML) with or without BCR-ABL1 translocation, and AML with BCR-ABL1 translocation.
4. HIV-positive patients and/or active HBV or HCV infection (as documented by positive HBV-DNA and HCV-RNA tests).
5. Clinically significant QTc prolongation (men > 450 ms; women > 470 ms), ventricular tachycardia, atrial fibrillation, second-degree heart block, history of myocardial infarction within the past year, congestive heart failure, and coronary artery disease requiring medication.
6. Active, uncontrolled severe infection.
7. History of other malignancies within the past 2 years, except for adequately treated in situ carcinoma of the cervix or breast; skin basal cell carcinoma or localized squamous cell carcinoma of the skin.
8. White blood cell count > 25 x 10^9/L. (This criterion can be met with hydroxyurea or leukapheresis.)
9. Mental impairment that would compromise the ability to participate in the study.
10. Any other situation in which the investigator believes that it would not be in the best interest of the patient to participate in the trial.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 24 months
  Defined as the highest dose at which less than 2 out of 6 (ie. 33%) participants experience a Dose-Limiting Toxicity (DLT).

SECONDARY OUTCOMES:
Complete Response Rate (CR) | Up to 24 months
  The percent of participants with morphologic complete remission (CR) according to modified International Working Group Acute Myeloid Leukemia Response Criteria (IWG AML)
Complete Response with incomplete blood count recovery (CRi) | Up to 24 months
  Meets all CR criteria, except for residual neutropenia < 1,000/µL or hrombocytopenia < 100,000/µL. Dependence on red blood cell (RBC) transfusions is also defined as CRi.
Disease free survival (DFS) | Up to 24 months
  Applies only to patients who achieve CR or CRi. It is measured from the date of remission to the date of relapse or death from any cause.
Overall survival (OS) | Up to 24 months
  Time from the start of the patient's initial treatment to the time of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Xu, Principal Investigator — The First Aiffiliated hosptical of xiamen University
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No